CLINICAL TRIAL: NCT01592383
Title: Phase II Study of Erlotinib for Patients With Malignant Peritoneal Mesothelioma (MPeM) Exhibiting EGFR Mutations
Brief Title: Erlotinib Hydrochloride in Treating Patients With Malignant Peritoneal Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0032; NCI-2012-00332 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Malignant Peritoneal Mesothelioma
MeSH Terms: interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive erlotinib hydrochloride PO QD. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774

SUMMARY:
The purpose of this study is to test the drug erlotinib (erlotinib hydrochloride) in people with malignant peritoneal mesothelioma who have a specific genetic mutation in their cancer. Erlotinib has been approved by the United States Food and Drug Administration (FDA) for other cancers, but erlotinib has not been approved for malignant peritoneal mesothelioma. This research is being done because there is no current standard treatment for malignant peritoneal mesothelioma and the study doctors want to see how erlotinib affects malignant peritoneal mesothelioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate (complete response [CR] + partial response [PR]) of erlotinib in malignant peritoneal mesothelioma (MPeM) patients who have epidermal growth factor receptor (EGFR) mutations.

SECONDARY OBJECTIVES:

I. To determine the percentage of patients with MPeM who have EGFR mutations. II. To characterize asbestos exposure history and other clinical parameters of patients with MPeM who do or do not have EGFR mutations.

III. To determine the disease control rate (CR + PR + stable disease [SD]) of MPeM patients who have EGFR mutations and are treated with erlotinib.

IV. To determine the progression-free survival (PFS) of MPeM patients who have EGFR mutations and are treated with erlotinib.

V. To determine the median overall survival (OS) of MPeM patients who have EGFR mutations and are treated with erlotinib.

VI. To evaluate toxicity in MPeM patients who have EGFR mutations and are treated with erlotinib.

TERTIARY OBJECTIVES:

I. To characterize the specific EGFR mutations observed in MPeM patients. II. To correlate tumor markers (cancer antigen [CA] 125 and soluble mesothelin-related peptide [SMRP]) with response rate, PFS, and OS in MPeM patients treated with erlotinib.

III. To correlate immunohistochemical staining of EGFR, phosphorylated (p)-EGFR, MET (Metastasis), E-cadherin, vimentin, and CBL (Casitas B-lineage Lymphoma)with EGFR mutational status and, if present, particular EGFR mutation noted.

IV. To correlate immunohistochemical staining of EGFR, p-EGFR, MET, E-cadherin, vimentin, and CBL with response rate, PFS, and OS in MPeM patients treated with erlotinib.

OUTLINE:

Patients receive erlotinib hydrochloride orally (PO) once daily (QD). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed malignant peritoneal mesothelioma; epithelial, sarcomatoid, biphasic, or well-differentiated papillary subtypes are allowed.
* A tumor block or 10 unstained slides must be available for determining EGFR mutational status; only those patients who have a mutation of the EGFR tyrosine kinase domain will be able to enroll in this study.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan.
* No prior use of EGFR tyrosine kinase inhibitors or monoclonal antibodies; all other prior treatments are allowed if >= 4 weeks since treatment completed, including chemotherapy (systemic or intraperitoneal), radiation therapy, and/or surgery; there is no limit on the number of previous treatments allowed.
* Life expectancy of greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Leukocytes >= 2,000/mcL.
* Absolute neutrophil count >= 1,500/mcL.
* Platelets >= 100,000/mcL.
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional ULN.
* Creatinine =< 2 X institutional ULN OR creatinine clearance >= 30 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
* The effects of erlotinib on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed screening and treatment consent.

Exclusion Criteria:

* Chemotherapy, radiotherapy, or surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop. progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib.
* EGFR-mutation negative tumor tissue as determined by sequencing; if an individual tissue test result is inconclusive (unable to be determined), it will be considered negative for study eligibility purposes.
* History of previous malignancy excluding non-melanoma skin lesions and in-situ cervical cancer; patients with other malignancies are eligible if they have been disease free for >= 3 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because it is unknown if erlotinib poses a potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with erlotinib, breastfeeding should be discontinued if the mother is treated with erlotinib.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with erlotinib; in addition, these patients are at increased risk of lethal infections; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Inability to tolerate or absorb an oral medication due to any cause, including but not limited to malabsorption syndromes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective Response Rate is calculated according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Time Frame: 1 year
Population: The study was terminated early after the enrollment of two participants and the data were not collected.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

2. Secondary Outcome: PFS
Description: Progression free survival (PFS) defined as time from study enrollment until disease progression or death.
Time Frame: 1 year
Population: The study was terminated early after the enrollment of two participants and the data were not collected.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: OS
Description: Overall survival measured as the time from study enrollment until death.
Time Frame: 1 year
Population: The study was terminated early after the enrollment of two participants and the data were not collected.
Groups:
- Treatment (Enzyme Inhibitor Therapy): Patients receive erlotinib hydrochloride PO QD. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  erlotinib hydrochloride: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicity
Description: Toxicity is calculated in terms of adverse events per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) criteria version 4.0
Time Frame: 30 days from the last dose of study drug
Population: The study was terminated early after the enrollment of two participants and the data were not collected.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Disease Control Rate - SD + PR + CR
Description: Disease Control Rate - SD + PR + CR is calculated as the percentage of patients with either complete response (CR: disappearance of all target lesions), or with partial response (PR: at least 30% decrease in the sum of longest diameter of target lesions, taking as reference the baseline sum longest diameter of target lesions), or stable disease (SD: neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease of an increase of at least 20% in the sum of the longest diameter of the target lesions taking as reference the smallest sum of longest diameter recorded since the treatment started or the appearance of one or more new lesions).
Time Frame: 1 year
Population: The study was terminated early after the enrollment of two participants and the data were not collected.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: EGFR Mutations Percentage
Description: EGFR Mutations Percentage is calculated as the percentage of patients who have activating EGFR mutations among all screened patients.
Time Frame: Baseline
Population: The study was terminated early after the enrollment of two participants and the data were not collected.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: An expected mild skin rash
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) — An expected mild skin rash
Fatigue (General disorders) | 1 (2)
Constipation (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT01592383/Prot_SAP_000.pdf